CLINICAL TRIAL: NCT02904447
Title: Plantar Forces Mid-term After Hemiarthroplasty With HemiCap for Hallux Rigidus
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Pernille Henszelman Jørsboe, Reservelæge, Copenhagen University Hospital, Hvidovre
Other Study IDs: HEMICAP
Record Dates: First submitted 2016-07-19; First posted 2016-09-19 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Hallux Rigidus
Keywords: hemicap; hallux rigidus
MeSH Terms: conditions — Hallux Rigidus | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: x-ray and pedobar foot pressure mapping

SUMMARY:
The purpose of this study is to examine variabel pressure gradients of the 1st toe, 2-5th toes and the metatarsal distal caput in patients who have had surgery with a partial proximal hemiarthroplasty in the 1st metatarsalphalangeal joint (MTP) between 2006-2014.

Also, to examine these variables and compare them to the totalt range of motion and pain, to find out if the measured pedobar pressure can be used identify the well treated patient and the poorly treated patient.

The pedobar pressure gradients will be compared with a control group with healthy feet.

ELIGIBILITY:
Inclusion Criteria:

* patients who has hemicap 1. MTP joint.

Exclusion Criteria:

* patients who haad revision surgery, for example removal of hemicap and desis og 1. MTP joint.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient who has had an operation with proximal hemiarthroplasty (hemicap) 1st MTP proximal prosthetics 2006-2014 in Hvidovre Hospital, Glostrup Hospital or Hamlet-Aleris Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Plantar forces under the hallux and the forefoot in patients operated with a hemiCAP in the 1st MTPJ. | One examination for each patient, approximately 30 min.
  Plantar forces are measured under the hallux and the forefoot (plantar pressure (kPa), maximal force (N), and force/time (N/s)) is measured by the Emed foot pressure mapping system.

SECONDARY OUTCOMES:
Range of motion (degrees) | One examination for each patient, approximately 30 min.
  Unit: degrees. ROM of the hemicap operated 1st MTPJ
Level of pain | One examination for each patient, approximately 30 min.
  Visual analog scale, 1-10 of the hemicap operated foot

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided